CLINICAL TRIAL: NCT05104190
Title: Comparison of Different Methods of Controlling Pain During Debonding of Orthodontic Brackets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Kashif Iqbal, Dr. Kashif Iqbal (orthodontist), Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Orthodontic pain
Record Dates: First submitted 2021-08-04; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Analgesia; Orthodontic Appliance Complication
Keywords: Orthodontic pain
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- plastic wafers group (Experimental): In one arm/ group 1 (plastic wafers group), debonding was done by open mouth technique. All brackets were removed using same plier i.e. angled direct bracket remover. Figure pressure in the apical direction was applied concomitantly applied to stabilize each tooth. Loose cotton was used between thumb and tooth during debonding. Arch wires and ligatures were not removed during debonding.
  Patient pain score during procedure was measured using visual analogue scale ranging from zero to one hundred (0-100) In
  Interventions: Other: Stabilization of teeth during debonding using fingure pressure and elastic wafer
- finger pressure group (Experimental): In another arm/ group 2( finger pressure group) brackets were removed in the same way with the same debonding plier as in group 1 but soft acrylic sheets folded 4 times were placed between upper and lower dentition with the patient biting on this wafer. Wires and ligatures were left tied to brackets during debonding. After the procedure, patient was asked about pain using visual analogue scale.
  Interventions: Other: Stabilization of teeth during debonding using fingure pressure and elastic wafer

INTERVENTIONS:
Other: Stabilization of teeth during debonding using fingure pressure and elastic wafer — To control pain during debonding in one group , teeth were stabilized with finger pressure with cotton between finger and teeth and then debonding using open mouth technique was done. In second group teeth were stabilized using a plastic wafer between maxillary and mandibular teeth and then debonding was done using closed mouth technique. In order to reduce biasness, all of the patients were debonded with same plier and with wires still ligated to brackets. With the help of VAS, pain score was measured after debonding. A single operator performed complete procedure of debonding and pain recording.

SUMMARY:
Purpose of this study was to evaluate different methods of controlling pain during debonding

DETAILED DESCRIPTION:
Patients data was obtained from the Department of Orthodontics, Armed Forces Institute of Dentistry, Rawalpindi. One Hundred and ten patients were included in the study, which were divided into two groups, 55 patients in each group, based on method of controlling pain during debonding. To control pain during debonding in one group , teeth were stabilized with finger pressure with cotton between finger and teeth and then debonding using open mouth technique was done. In second group teeth were stabilized using a plastic wafer between maxillary and mandibular teeth and then debonding was done using closed mouth technique. In order to reduce biasness, all of the patients were debonded with same plier and with wires still ligated to brackets. With the help of VAS, pain score was measured after debonding. A single operator performed complete procedure of debonding and pain recording.

ELIGIBILITY:
Inclusion Criteria:

Patients between 13-21 years of age who can understand, assess, and answer the questionnaires. 2) No missing teeth except extracted premolars 3) Undergoing upper and lower fixed orthodontic treatment with Roth prescription 0.022-inch metal brackets . 4) Finishing arch wires present for at least two months

Exclusion Criteria:

1. The subjects with a previous history of facial or mandibular surgery or syndromes affecting the jaw or face .
2. Patient with history of jaw sugeries.
3. Patients with history of taking medicine periodically or in the last 24 hours (eg, painkillers, corticosteroids, and antiflu drugs),
4. Patient with history of debonded brackets and replacement.
5. Patient with history of tooth transplantation or microscrews placement.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 148 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Measurement of pain | Immediatey after debonding
  Using visual analogue scale pain was measured

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Khalid, BDS, FCPSII, Study Chair — AFID
Locations (1):
- Kashif Iqbal, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No